CLINICAL TRIAL: NCT01879982
Title: A Personal Wearable and Interactive System for Monitoring and Multivariable Physiological Assessment to Predict Mood Changes: a Pilot Study With Cyclothymic and Rapid Cycling Bipolar Subjects
Brief Title: PSYCHE (Personalised Monitoring SYstems for Care in Mental Health)
Acronym: PSYCHE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A00725-38
Record Dates: First submitted 2013-03-22; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Disorder I; Bipolar Disorder II; Rapid Cycling Bipolar Disorder(DSM-IV-TR)
Keywords: Bipolar disorder; subtypes
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wellness Wearable System & Smartphone

SUMMARY:
For the moment, the detection of a mood episode in Bipolar Disorder (BD) relies on the appearance of the first clinical signs that the clinician detect or that the patient becomes aware of and reports to the clinician. Since physiological parameters such as cardiac rhythms, respiratory rate, voice characteristics and actigraphy seem to be related to the onset of a mood episode, information collected through the combined monitoring of multiple selected physiological parameters (such as cardiac rhythms, respiratory rate, movements, voice) during wake and sleep time, using wearable user friendly systems included into garments as well as with a smartphone, may offer a new perspective in the long-term treatment of BD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals aged from 18 to 65 years old (both ages included).
2. Participants meeting DSM-IV-TR criteria for bipolar disorder I or II subtypes or Participants meeting DSM-IV-TR criteria for rapid cycling BD, which is defined by a pattern of presentation accompanied by 4 or more mood episodes in a 12-month period, with a typical course of mania or hypomania followed by depression or vice versa. The episodes must be demarcated by a full or partial remission lasting at least 2 months or by a switch to a mood state of opposite polarity.
3. Female participants must agree to use efficient contraceptive methods during the study duration.
4. Participants must have signed informed consent documents indicating that they understand the purpose and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions.
5. Patients must be affiliated with or a beneficiary of a social security system.

Exclusion Criteria:

1. Any clinically relevant acute or chronic diseases which could interfere with the participants' safety during the trial, or expose them to undue risk or which could interfere with the study objective. This last perspective includes :- Attention deficit and hyperactivity disorder (ADHD)- Borderline personality disorder (BPD)
2. Current MDD episode or manic episode, according to the DSM-IV-TR criteria
3. Current major suicidal ideation (suicidal thoughts several times a day)
4. History of recent (less than 1 year preceding inclusion) substance abuse or dependence (tobacco dependence excepted)
5. Pregnant women as determined by the patient or breast-feeding women
6. Any history of significant allergy.
7. No legal capacity or limited legal capacity or unable to give an informed consent.
8. Participants unlikely to co-operate in the study, and/or poor compliance anticipated by the investigator
9. Participants being in the exclusion period according to the French National File for participants participating in a biomedical research.
10. Total annual amount of compensation earned from participating in clinical studies exceeding 4500 Euros.
11. Patients with pacemaker, defibrillator, or any implanted electronic device (to avoid any hazard - see section 7.3.2 of the Psyche device User Manual).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cyclothymia or with rapid cycling BD will be recruited in the general population via ads in newspapers and universities (psychology, medical, and arts departments, for instance) and in clinical populations (patients from the investigators).
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
detect and predict mood changes in cyclothymic subjects and in rapid cycling subjects | 14-week study assessment
  recording heart rate, respiratory rate and body activity with a wearable device ("Wearable Wellness System" or WWS), and by analysing subject's voice through a voice analysis system embedded in a smartphone.

SECONDARY OUTCOMES:
tolerability and acceptability of the regular use of PSYCHE multiparameter platform (WWS and the smartphone)and the feasibility and the different functionalities of the different components of the PSYCHE system in a field trial | 14-week assessment study
  Evaluation criteria will be :
  1. Subjective : the proportions of subjects with tolerance problems and with acceptance of future use, for the different components of the system, as assessed with the end-of-study criteria or as reported at the end of the visits on the basis of an open question ;
  2. Objective: the proportion of missing appointments (daily and biweekly recordings) . Evaluation criteria will be :
  1) Subjective : the proportions of subjects with tolerance problems and with acceptance of future use, for the different components of the system, as assessed with the end-of-study criteria or as reported at the end of the visits on the basis of an open question ; 2) Objective: the proportion of missing appointments (daily and biweekly recordings) 3) Evaluation criteria will be the estimated frequencies and types of technical and professional user problems during the study (according to a qualitative methodology)

CONTACTS AND LOCATIONS:
Overall Officials: Bertschy Gilles, MD, Principal Investigator — Service de Psychiatrie II - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Psychiatrie II - Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France